CLINICAL TRIAL: NCT07304908
Title: Perception-based Interventions Affect Public Acceptance of Using Large Language Models in Medicine: Randomized Controlled Trial
Brief Title: Effect of Perception-based Interventions on Public Acceptance of Using Large Language Models in Medicine
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Liu Jue, Prof., Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NNSF72474005
Record Dates: First submitted 2025-12-01; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Large Language Models; Acceptability of Health Care; Perception, Self
Keywords: Large language model; Artificial intelligence; Perception-based interventions; Public acceptance
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Perceived benefits of large language models in medicine (Experimental): Participants were asked to read "In April 2023, Massachusetts General Hospital launched a pilot program utilizing medical LLMs to assist with emergency department triage and initial diagnosis and observed a reduction in patient wait times and an improvement in clinical efficiency."
  Interventions: Other: Perception-based interventions
- Perceived racial bias in large language models in medicine (Experimental): Participants were asked to read "In November 2022, a research team from the University of California, San Francisco found that cutting-edge medical LLMs exhibited racial bias when recommending treatment plans."
  Interventions: Other: Perception-based interventions
- Perceived ethical conflicts in large language models in medicine (Experimental): Participants were required to read "In February 2023, a major European hospital network inadvertently leaked partially anonymized but still sensitive patient data during the testing of medical LLMs due to a system configuration error. Although no direct patient harm occurred, this increased public concerns regarding data privacy and security and compelled relevant institutions to conduct urgent reviews of their data protection measures."
  Interventions: Other: Perception-based interventions
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Perception-based interventions — Participants allocated to the intervention group received perception-based interventions. Interventions for Groups 1-3 were perceived benefits of LLMs in medicine, perceived racial bias in LLMs in medicine, and perceived ethical conflicts in LLMs in medicine, respectively.
  Arms: Perceived benefits of large language models in medicine; Perceived ethical conflicts in large language models in medicine; Perceived racial bias in large language models in medicine

SUMMARY:
Large language models (LLMs) show promise in medicine, but concerns about their accuracy, coherence, transparency, and ethics remain. To date, public perceptions on using LLMs in medicine and whether they play a role in the acceptability of health care applications of LLMs are not yet fully understood. This study aims to investigate public perceptions on using LLMs in medicine and if interventions for perceptions affect the acceptability of health care applications of LLMs.

DETAILED DESCRIPTION:
Owing to rapid advances in artificial intelligence, large language models (LLMs) are increasingly being used in a variety of clinical settings such as triage, disease diagnosis, treatment planning, and self-monitoring. Despite their potential, the use of LLMs remains restricted within healthcare settings due to lack of accuracy, coherence, and transparency and ethical concerns. Public perceptions such as perceived usefulness and risks play a crucial role in shaping their attitudes towards artificial intelligence that can either facilitate or hinder its adoption. Yet, to our knowledge, there is lack of awareness about perception-driven interventions in health care and no previous studies have examined whether public perceptions play a role in the acceptability of medical applications of LLMs. Hence, this study aims to investigate public perceptions on using LLMs in medicine and if interventions for perceptions affect the acceptability of health care applications of LLMs.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Capable of completing an online survey
* Agree to sign an informed consent form

Exclusion Criteria:

* Unable to answer questions or communicate
* Not willing to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who will change their attitudes towards medical applications of large language models | Through study completion, an average of 1 year
  Public acceptance of applying large language models to medicine will be categorized into yes, not sure, and no, which will be collected before perception-based interventions and after interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Jue Liu, Principal Investigator — Peking University
Locations (1):
- Jue Liu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No